CLINICAL TRIAL: NCT03075475
Title: Study of Effectiveness of a Treatment to Improve the Mental Health of Children and Adolescents Affected by Armed Conflict in Kachin State, Myanmar
Brief Title: Effectiveness Study of a Treatment to Improve the Mental Health of Children and Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very few children and adolescents identified who met intake criteria.
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00007317
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Child Mental Disorder; Behavior Problem
Keywords: Child; Adolescent; Mental Health; Randomized Controlled Trial
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CETA Treatment (Experimental): For treatment group participants, they will then have weekly Common Elements Treatment Approach (CETA) counseling sessions with a counselor lasting no more than 1.5 hours per session, and a total of approximately 10-12 sessions. They will then repeat the assessment instrument after their last session, as well as 6 months after finishing treatment, and these meetings will again last no more than 1.5 hours. All total, it is expected that treatment group participants will have 13 meetings with a study team member or counselor over the course of their participation.
  Interventions: Behavioral: Common Elements Treatment Approach
- Waitlist (No Intervention): Waitlist group participants be contacted by a study team member from the local partner organization regularly (weekly) while they are on the wait list. These contacts from the study team will be short and last less than 30 minutes and will be used to briefly assess symptom levels and safety. At the end of their wait period, they will be asked to complete the assessment instrument a second time and this meeting will take no more than 1.5 hours. For participants in the waitlist group, we estimate 13 meetings total during their wait period (2 meetings of no more than 1.5 hours, 10 contacts less than 30 minutes).

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach — The Common Elements Treatment Approach (CETA), is a trans-diagnostic psychotherapy that is based on common evidence-based treatments for depression, anxiety, trauma and stress related disorders. This treatment can be used to treat individuals with any of these mental health problems and with any combination of these problems. CETA expands upon traditional treatment approaches that are designed to focus on one specific disorder and has been proven through multiple rigorous trials to reduce the burden of multiple common mental health problems and improve functionality among men and women living in low resource settings. CETA can be provided to people in their own communities by trained and supervised lay providers, for example community health workers.
  Other Names: CETA
  Arms: CETA Treatment

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a psychotherapeutic intervention, the Common Elements Treatment Approach (CETA), to address the mental health needs of children and adolescents age 8-17 who have been affected by armed conflict in Kachin State, Myanmar. The 10-12 week talk-based counseling treatment, delivered by community mental health workers, will be evaluated against a wait-list control group. This project follows on a recently completed trial of CETA for adult trauma survivors from Myanmar along the Thai-Myanmar border which found that CETA was acceptable, accessible, and effective in improving mental health and functioning of adults. The investigators hypothesize that the intervention will be similarly effective for improving the mental health and functioning of children and adolescents.

DETAILED DESCRIPTION:
The Common Elements Treatment Approach (CETA) is a trans-diagnostic psychotherapeutic intervention.

Results from qualitative interviews following the randomized controlled trial (RCT) of CETA for adults (IRB # 00003601) and during the scale-up of CETA services have indicated that there is a major need for mental health services for children and adolescents in Myanmar, as currently there are no evidence-based psychotherapy services for children and adolescents in the country. Specifically, since the initial trial the research team has received requests from community-based organizations to implement CETA for children and adolescents in Kachin language-speaking communities in northern Myanmar. Local partners and the Applied Mental Health Research group (AMHR) at Johns Hopkins University (JHU) believe that CETA is amenable for use with children and adolescents and that this population would benefit in similar ways to adults. A qualitative study has since been conducted (IRB# 00006933), and the data used to develop and validate an assessment instrument with children and adolescents in Kachin state (IRB# 00006929).

The JHU research team will work with the local partner organization, Kachin Baptist Convention (KBC), to implement this project. KBC is a well-established community-based organization that currently provides emergency relief services to approximately 20,000 displaced Kachin people living in 42 camps. Their community outreach activities are non-denominational.

Participants will mostly be accessed through schools and in partnership with the local implementing partner. Their teachers, secondary caregivers and persons from the local partner organization who work with them regularly - all of whom are involved in the study as key community informants - will identify and refer the potential child/adolescent participants for screening into the study. Screening will otherwise be open to all children/adolescents, and those who are eligible will be asked to participate in the trial. Informed consent will be obtained from the parent/guardian and informed assent from the child. Participants will be randomly assigned to either receive CETA immediately or be put on a waitlist to receive treatment later.

Counselors will be current employees of the local partner organization who have participated in a 2-week initial training followed by 8-10 weeks of supervised practice. Counselors will receive weekly clinical supervision for the duration of the trial.

During the RCT, 10-12 weekly CETA sessions will be delivered individually in private spaces either at schools, homes, or in the community. In most cases, the children are living in the camps with their parents/guardians. Counselors will also follow-up with control children on a weekly basis to assess their symptoms using a client monitoring form. Both treatment and control participants will be reassessed using the same assessment instrument following the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Moderately or severely affected (cutoff to be defined during validation phase) children ages 8-17 years.

Exclusion Criteria:

* Active psychosis or serious developmental disorder (e.g., mental retardation, autism) that would preclude participation in cognitive-behavioral oriented skills intervention

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Change in child mental health scores from composite measure | The time between pre- and post-test intervention assessment will be 8-12 weeks for treatment group (according to the number of CETA sessions) and 10 weeks for wait list participants.
  Self-reported child mental health symptoms will be measured using a modified, locally validated version of the assessment instrument consisting of 23 items from 1) the Child PTSD Symptom Scale (CPSS); 2) and the Moods and Feelings Questionnaire (MFQ); and 3) items developed from qualitative research in this population. Respondents report how often each problem has bothered him/her in the past two weeks. Response options range from 0 "none of the time" to 3 "almost all of the time". Results will be reported as a single value from this composite outcome measure consisting of multiple measures.

SECONDARY OUTCOMES:
Change in child behavior problem scores | The time between pre- and post-test intervention assessment will be 8-12 weeks for treatment group (according to the number of CETA sessions) and 10 weeks for wait list participants.
  Self-reported child behavior problems will be assessed using a behavior problem checklist developed using qualitative data collected from this population. Respondents report how often they have done or experienced each behavior in the past two weeks. Response options range from 0 "none of the time" to 3 "almost all of the time".
Change in child functional impairment | The time between pre- and post-test intervention assessment will be 8-12 weeks for treatment group (according to the number of CETA sessions) and 10 weeks for wait list participants.
  Self-reported child functional impairment will be assessed using a functioning scale developed using qualitative data collected from this population. Respondents report how much difficulty they currently have doing tasks of daily living. Response options range from 0 "no difficulty" to 3 "often cannot do".

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lee, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Kachin Baptist Convention Jan Mai Kawng Camp, Myitkyina, Kachin State, Burma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolton P, Lee C, Haroz EE, Murray L, Dorsey S, Robinson C, Ugueto AM, Bass J. A transdiagnostic community-based mental health treatment for comorbid disorders: development and outcomes of a randomized controlled trial among Burmese refugees in Thailand. PLoS Med. 2014 Nov 11;11(11):e1001757. doi: 10.1371/journal.pmed.1001757. eCollection 2014 Nov. PMID 25386945